CLINICAL TRIAL: NCT02770586
Title: Comparison of Positron Emission Mammography and Contrast-enhanced Breast MRI in Women With a High Suspicion of Breast Cancer
Brief Title: Comparison of Positron Emission Mammography and Contrast-enhanced Breast MRI
Acronym: PEM/MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15-004872
Record Dates: First submitted 2016-02-17; First posted 2016-05-12 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breast PET (Other): Breast PET
  Interventions: Diagnostic Test: Breast PET

INTERVENTIONS:
Diagnostic Test: Breast PET — imaging of the breast using the Breast PET system

SUMMARY:
The hypothesis of this study is that positron emission mammography will provide comparable sensitivity to contrast-enhanced breast MRI in women with a high suspicion of breast cancer.

The aim of this study is to determine the sensitivity of Positron Emission Mammography (PEM) relative to that of Contrast-enhanced breast MRI (CE-MRI) in women with a high suspicion of breast cancer

DETAILED DESCRIPTION:
Study Overview:

The study population will comprise 150 women with a BI-RAD 5 or 6 finding on recent imaging who are scheduled for contrast enhanced breast MRI. Recruitment will be from the pool of patients scheduled for an MRI in the Department of Radiology at Mayo Clinic Rochester. All patients will have a PEM study within 5 business days of the clinically indicated MRI. Subjects must meet the following eligibility criteria:

1. Recent imaging study (mammogram, tomosynthesis, MBI or ultrasound) interpreted as highly suggestive of malignancy or a known biopsy proven malignancy [Breast Imaging Reporting and Data System (BI-RADS) Category 5 or 6]
2. Scheduled to undergo or has recently undergone a contrast-enhanced breast MRI
3. Age 25 or older

The interpretation will be performed by different study radiologists blinded to the results of the other study. Prior breast imaging studies (mammography, tomosynthesis, MBI and ultrasound) and medical record will be available to the interpreting physician. Following the separate interpretations, an integrated interpretation of the MRI and PEM images will be performed to match any lesions seen and determine final clinical management of the patient.

Reference standard will be surgical pathology or biopsy. For findings that were not resolved through biopsy or surgery, follow up data, including any imaging and / or biopsies performed in the 365 day period following study entry (date of the study PEM) will be collected through medical record review (and patient interview for those who do not return for further clinical management).

The primary analysis is to compare the PEM diagnostic yield to the MRI diagnostic yield, which is considered the standard for this trial. The primary analysis will use the observed MRI diagnostic yield as the control value.

If the 95% Confidence Interval (CI) for the PEM diagnostic yield lies entirely below the MRI diagnostic yield value, PEM will be deemed inferior to MRI for detecting breast cancer in this patient population. If the 95% CI for the PEM diagnostic yield contains the MRI diagnostic yield value, PEM will be deemed equivalent to MRI for detecting breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* All women in this study will have recent imaging study (mammogram, tomosynthesis, MBI or ultrasound) interpreted as highly suspicious for malignancy or known biopsy-proven malignancy (BI-RADS Category 5 or 6 within 60 days prior to the MRI or PEM study
* Scheduled or will be scheduled for clinically indicated contrast-enhanced breast MRI examination
* PEM must be performed within 5 business days, prior to or following the clinical MRI
* Participant has signed the study-specific informed consent prior to registration
* Age 25 or older

Exclusion Criteria:

* Unable to understand and sign the consent form
* Pregnant or lactating
* Physically unable to lie prone for ~20 minutes
* Undergone bilateral mastectomy
* Weight more than 300 lbs (weight limit on PEM table)
* Have contraindications to the clinical MRI examination
* Scheduled to undergo breast biopsy or surgery in the time period between the PEM and MRI studies

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-08; Primary Completion 2019-06-11 (Actual); Study Completion 2019-10-12 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield of breast cancers detected on PEM compared to MRI | One week
  The primary analysis is to compare the PEM diagnostic yield to the MRI diagnostic yield, which is considered the standard for this trial. The primary analysis will use the observed MRI diagnostic yield as the control value. The diagnostic yield of PEM will be estimated with a binomial point estimate and corresponding 95% binomial confidence interval (CI). The point estimate for the diagnostic yield (for both MRI and PEM) will be the number of confirmed breast cancers detected by the imaging (i.e. as determined by the reference standard) divided by the number of eligible and evaluable patients.

CONTACTS AND LOCATIONS:
Overall Officials: Michael O'Connor, PHD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials